CLINICAL TRIAL: NCT05635422
Title: Pilot Study to Evaluate an Isokinetic Fatigue Index for Prevention Purposes in a Population of Triathletes
Brief Title: Isokinetic Fatigue Index in a Population of Triathletes
Acronym: ISOTRIFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boulogne sur Mer Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-01
Record Dates: First submitted 2022-11-15; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- isokinetism test in high level triathletes practicing an endurance sport (Experimental)
  Interventions: Diagnostic Test: isokinetism test

INTERVENTIONS:
Diagnostic Test: isokinetism test — measure of muscular fatigability by isokinetism

SUMMARY:
The aim of this study is to evaluate the relevance of carrying out a measure of muscular fatigability by isokinetism, in the search for factors favouring micro-traumatic lesions of the lower limbs in a population of triathletes.

This is a prospective monocentric pilot study of the before/after type in which the patient is his or her own control, in high-level triathletes practising an endurance sport, who have had more than 7 consecutive days off running due to a musculoskeletal injury during the previous sporting year.

ELIGIBILITY:
Inclusion Criteria:

* Having had a practical running break of more than 7 consecutive days due to a musculoskeletal injury of a lower limb during the previous sport year
* Willing to comply with all study procedures
* Having given written consent
* Socially insured

Exclusion Criteria:

* Pain that does not allow an isokinetic test to be performed
* Knee joint amplitude less than 100° of flexion or flessum greater than 5°.
* History of rupture or ligamentoplasty of the anterior cruciate ligament less than 2 years ago
* History of knee surgery less than 2 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
fatigue index between the injured leg and the healthy leg | the day of inclusion
  To compare the fatigue index between the injured leg and the healthy leg in high level triathletes injured in the previous season.

SECONDARY OUTCOMES:
difference of the fatigue index to the difference of the Croisier ratio between the injured leg and the healthy leg | the day of inclusion
  Correlate the difference in the fatigue index to the difference in the Croisier ratio between the injured leg and the healthy leg.

CONTACTS AND LOCATIONS:
Locations (1):
- Boulogne sur mer Hospital Center, Boulogne-sur-Mer, France